CLINICAL TRIAL: NCT05633121
Title: Retrospective Study Evaluating the Contribution of Rheopheresis in the Treatment of Uremic Calciphylaxis
Brief Title: Retrospective Study Evaluating the Contribution of Rheopheresis in the Treatment of Uremic Calciphylaxis (RHEO-CUA)
Acronym: RHEO-CUA
Status: Completed | Type: Observational
Sponsor: Association ECHO (Other)
Collaborators: European Clinical Trial Experts Network (Other); Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: RHEO-CUA
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Rheopheresis; Calcifying Uremic Arteriolopathy; Uremic Calciphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient suffering from uremic calciphylaxis treated with rheopheresis
  Interventions: Procedure: Rheopheresis
- Patient suffering from uremic calciphylaxis not treated with rheopheresis

INTERVENTIONS:
Procedure: Rheopheresis — Technique of apheresis in double filtration, allowing the extraction of molecules of high molecular weight, and thus the improvement of the rheological conditions of microcirculation. The expected effect is the improvement of tissue oxygenation and the acceleration of the healing of skin lesions, with the consequent reduction of infectious complications.
  Groups: Patient suffering from uremic calciphylaxis treated with rheopheresis

SUMMARY:
Calcifying uremic arteriolopathy (or uremic calciphylaxis) is a rare disease (prevalence <1% of dialysis patients), but the prognosis is often catastrophic. The main non-modifiable risk factors are age, female gender, diabetes, obesity and length of time on dialysis. Today, there is no specific treatment for this pathology, and the therapeutic management is poorly codified. However, it is commonly accepted that the treatment is based on the control of risk factors, local care, and the possible addition of treatment with sodium thiosulfate. Hyperbaric oxygen therapy has also been proposed by some authors, but remains not very accessible in practice.

Recently, it has been proposed to use Rheopheresis as an adjuvant treatment for severe forms of uraemic calciphylaxis. It is a technique of apheresis in double filtration, allowing the extraction of molecules of high molecular weight, and thus the improvement of the rheological conditions of microcirculation. The expected effect is the improvement of tissue oxygenation and the acceleration of the healing of skin lesions, with the consequent reduction of infectious complications.

The aim of this study is to propose a large national retrospective study, studying the evolution of patients with uremic calciphylaxis and treated by rheopheresis, compared to a control group. This will allow to have a more precise idea of the contribution of Rheopheresis in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Chronic hemodialysis
* Uraemic calciphylaxis (clinical or histological diagnosis) diagnosed between January 2010 and December 2022,
* Rheopheresis treatment initiated within one month of calciphylaxis diagnosis (for the exposed group)
* Patient informed and not opposed to the use of their health data.

Exclusion Criteria:

* minor patient,
* Advanced cognitive disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient on chronic hemodialysis and suffering from uraemic calciphylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients fully recovered 6 months after diagnosis. | 6 months
  Complete healing will be defined by the healing of all skin lesions without the appearance of new ones.

CONTACTS AND LOCATIONS:
Locations (1):
- ECHO - Pole Santé Sud, Le Mans, France